CLINICAL TRIAL: NCT07075601
Title: Non-interventional Study Exploring the Composition of the Valvular Microbiota of Patients Undergoing Cardiac Surgery
Acronym: BIOVALV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/25/0020; 2025-A00422-47 (Other: N°ID-RCB number)
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Valvulopathy; Cardiac Surgery; Microbiota
MeSH Terms: conditions — Heart Valve Diseases | interventions — Blood Specimen Collection; Sequence Analysis, DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with an indication for cardiac surgery (Experimental): Patients with an indication for cardiac surgery during which the aortic valve is explanted.
  Interventions: Biological: Take 1 ml of blood; Biological: DNA sequencing; Procedure: Valve collection (healthcare waste); Other: Collection of serious post-operative complications

INTERVENTIONS:
Biological: Take 1 ml of blood — Take 1 ml of blood
Biological: DNA sequencing — DNA sequencing
Procedure: Valve collection (healthcare waste) — Valve collection (healthcare waste)
Other: Collection of serious post-operative complications — Collection of serious post-operative complications

SUMMARY:
The prevalence of aortic valve disease is increasing, with these valvulopathies present in half of individuals over the age of 65.

Oberbach A. et al (1) demonstrated the presence of microbiota in 52% of cases of explanted aortic valves. One current hypothesis is the role of this microbiota in the pathophysiology of these degenerative valve diseases. This microbiota is probably not completely eradicated after resection of the native valve and implantation of a conventional prosthesis; it is even left in place during percutaneous aortic valve implantation, during which the prosthesis is deployed within the native valve. It could therefore also play a role in the occurrence of postoperative complications and the degeneration or thrombosis of a bioprosthesis.

Furthermore, recent clinical and epidemiological studies have shown a link between oral infections and cardiovascular diseases. As recommended by the HAS, these patients require multidisciplinary care, involving cardiologists, cardiac surgeons and general practitioners, as well as careful oral and dental care and monitoring provided by specialists in oral pathologies and oral care. The accumulation of bacterial plaque on the surface of the tooth and certain oral bacteria causes the development of periodontal pockets which are characteristic of periodontitis. Bacteria, microbial products and inflammatory mediators produced locally can then enter the bloodstream and affect distant organs such as the cardiovascular system. The recommendations of the European Society of Cardiology are therefore to carry out regular oral and dental consultations to prevent the risk of infection. Therefore, within the Toulouse University Hospital, a care network has been set up for patients with cardiovascular pathologies, in order to improve their access to dental care, screening and management of oral diseases. For the past year, patients hospitalized in the cardiology departments have been seen in consultation in the dental department of the Toulouse University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient.
* Present an indication for cardiac surgery that requires explantation of the aortic valve.
* Be able to receive information about the study process and understand the study participation information form.
* State their non-opposition to participating in the study.

Exclusion Criteria:

* Patients infected with HIV
* Age under 18
* Under court supervision, guardianship, or curatorship
* Patients with a history of infective endocarditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a serious postoperative complication | 48 months
  Number of ischemic or hemorrhagic strokes; re-intervention, infective endocarditis, aortic bioprosthesis degeneration, aortic bioprosthesis thrombosis, mortality, surgical site infection requiring repeat surgery

SECONDARY OUTCOMES:
Determine the microbiological composition of saliva | 48 months
  Determine the components of the salivary microbiota
Determine the components of the microbiota of periodontal plaque | 48 months
  Determine the components of the microbiota of periodontal plaque
Oral health assessment | 48 months
  Oral health assessment using the oral health assessment questionnaire called "Oral Study" which asks questions about the use of a toothbrush, interdental brushes, the frequency of visits to the dentist, and the use of mouthwash.
Evaluation of hygiene and dietary habits | 48 months
  Assessment of dietary habits using a questionnaire on eating habits and the frequency of consumption of certain foods (bread, rusks, rice, pasta, vegetables, fruits, dairy products, fish, meat) with multiple choices between:
  Several times a day - Once a day - Several times a week - Once or twice a month - Never
Determine the inflammatory composition of saliva | 48 months
  Determining inflammatory molecules in saliva
Determine the immune composition of saliva | 48 months
  Determine the immune cells and molecules found in saliva
Determine the microbiological composition of feces | 48 months
  Determine the molecules that make up the fecal microbiota

CONTACTS AND LOCATIONS:
Locations (1):
- Rangueil Hospital, Toulouse, France, France

IPD SHARING:
Plan to Share IPD: No